CLINICAL TRIAL: NCT00120458
Title: Black Cohosh Therapy for Menopause-Related Anxiety
Brief Title: Black Cohosh as Alternative Therapy for Treating Menopause-Related Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Jay D. Amsterdam, M.D., University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT002289-01A1 (NIH); R21AT002289-01A1 (NIH)
Record Dates: First submitted 2005-07-14; First posted 2005-07-18 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Generalized Anxiety Disorder; Menopause
Keywords: Black Cohosh; Cimicifuga; Anxiety; Women; Complementary and Alternative Medicine
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Anxiolytic Therapy
  Interventions: Dietary Supplement: Black cohosh
- 2 (Placebo Comparator): Anxiolytic Therapy
  Interventions: Dietary Supplement: Black cohosh

INTERVENTIONS:
Dietary Supplement: Black cohosh — 32 to 128 mg (black cohosh)
  1 to 4 capsules daily (placebo)

SUMMARY:
This study will determine the effectiveness of the herb black cohosh for treating menopause-related anxiety symptoms in women.

Study hypotheses: 1) Black cohosh will have a superior anti-anxiety effect compared to placebo. 2) Black cohosh will have a comparable safety profile to that of placebo.

DETAILED DESCRIPTION:
During menopause, up to 90% of women will experience symptoms of anxiety, such as nervousness, irritability, fatigue, muscle aches, depression, and low libido. Concern over the safety and effectiveness of hormone replacement therapy for relieving these symptoms has caused many women to seek alternative medical treatments. Data suggest that black cohosh has a direct effect on the neurotransmitters and receptors involved in anxiety. This study will determine whether black cohosh can effectively treat anxiety symptoms in menopausal women.

This study will last 12 weeks. Participants will be randomly assigned to receive either black cohosh or placebo daily for the duration of the study. Self-report scales will be used to assess participants' anxiety symptoms and quality of life at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing menopause or postmenopausal
* Have symptoms of menopause-related anxiety

Exclusion Criteria:

* Any form of generalized anxiety disorder (GAD) unrelated to menopause
* Onset of GAD at least 3 years prior to menopause or at least 5 years after menstruation has stopped
* Alcohol or drug dependence within 3 months prior to study entry
* Allergy to black cohosh
* History of hormone replacement therapy
* Current use of vaginal estrogen cream or phytoestrogens
* Current use of tranquilizers, antidepressants, or antianxiety therapies
* Abnormal uterine bleeding
* History of estrogen-dependent cancer
* History of endometrial hyperplasia (abnormal increase in cells) or endometrial cancer
* Rapidly growing uterine fibroids
* Abnormal finding upon gynecological examination that would interfere with the study
* Abnormal breast examination or mammogram
* Any unstable medical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Score on Hamilton Anxiety Rating Scale | 12 Weeks

SECONDARY OUTCOMES:
Quality of life and functional outcome ratings | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay D. Amsterdam, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Amsterdam JD, Yao Y, Mao JJ, Soeller I, Rockwell K, Shults J. Randomized, double-blind, placebo-controlled trial of Cimicifuga racemosa (black cohosh) in women with anxiety disorder due to menopause. J Clin Psychopharmacol. 2009 Oct;29(5):478-83. doi: 10.1097/JCP.0b013e3181b2abf2. PMID 19745648